CLINICAL TRIAL: NCT00740779
Title: A Multi-Center, Double-Blind, Placebo-Controlled Investigation of Silodosin in the Treatment of Subjects With Moderate to Severe Abacterial Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Brief Title: Use of Silodosin to Treat Moderate to Severe Abacterial Chronic Prostatitis/Chronic Pelvic Pain Syndrome.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SI08001
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-01

CONDITIONS: Abacterial Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Keywords: prostatitis, chronic pelvic pain
MeSH Terms: conditions — Prostatitis | interventions — silodosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Silodosin 4 mg (Experimental): 4 mg daily
  Interventions: Drug: Silodosin 4 mg
- Silodosin 8 mg (Experimental): Silodosin 8 mg daily
  Interventions: Drug: Silodosin 8 mg
- Placebo (Placebo Comparator): 1 placebo capsule daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silodosin 8 mg — Silodosin 8 mg daily
  Other Names: Rapaflo
  Arms: Silodosin 8 mg
Drug: Placebo — Placebo
  Other Names: Placebo control.
  Arms: Placebo
Drug: Silodosin 4 mg — Silodosin 4 mg daily
  Other Names: Rapaflo
  Arms: Silodosin 4 mg

SUMMARY:
The primary objective is to compare the efficacy of silodosin 4 and 8 mg once daily with placebo in the treatment of subjects with moderate to severe abacterial chronic prostatitis/chronic pelvic pain syndrome during a 12 week treatment period. The secondary objective is to compare the safety of silodosin 4 and 8 mg once daily with placebo.

DETAILED DESCRIPTION:
A Multi-Center, Double-Blind, Placebo-Controlled Investigation of Silodosin in the Treatment of Subjects With Moderate to Severe Abacterial Chronic Prostatitis/Chronic Pelvic Pain Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male, at least 18 years of age
* Has a total NIH-CPSI total score of 15
* Has a NIH-CPSI pain score of 8
* Has had pain in the pelvic region for at least 3 months prior to screening

Exclusion Criteria:

* Has previously participated in a Watson study with silodosin
* Has previously received α-blocked therapy for chronic prostatitis/chronic pelvic pain syndrome or is currently receiving α-blocked therapy for any condition
* Has experience ≥2 urinary tract infections within the previous 12 months
* Has any medical condition that in the opinion of the investigator precludes safe participation in the study
* Has any medical condition that could confound the efficacy evaluation
* Is receiving ketoconazole, or other known potent inhibitors of cytochrome P450 3A4 or any medication in the opinion of the investigator that precludes safe participation in the study
* Is receiving any medication that in the opinion of the investigator that could confound the efficacy evaluation
* Has participated in a study involving the administration of an investigational agent within the past 30 days

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Caramelli, MS, Study Director — Watson Pharmaceuticals
Locations (22):
- United States (22):
  - Watson Investigational Site, San Diego, California
  - Watson Investigational Site, Denver, Colorado
  - Watson Investigational Site, Columbus, Georgia
  - Watson Investigational Site, Roswell, Georgia
  - Watson Investigational Site, Jeffersonville, Indiana
  - Watson Investigational Site, West Des Moines, Iowa
  - Watson Investigational Site, Baltimore, Maryland
  - Watson Investigational Site, Boston, Massachusetts
  - Watson Investigational Site, Watertown, Massachusetts
  - Watson Investigational Site, Omaha, Nebraska
  - Watson Investigational Site, Voorhees Township, New Jersey
  - Watson Investigational Site, Albuquerque, New Mexico
  - Watson Investigational Site, Garden City, New York
  - Watson Investigational Site, Kingston, New York
  - Watson Investigational Site, New York, New York
  - Watson Investigational Site, Poughkeepsie, New York
  - Watson Investigational Site, Columbus, Ohio
  - Watson Investigational Site, Bethany, Oklahoma
  - Watson Investigational Site, Edmond, Oklahoma
  - Watson Investigational Site, State College, Pennsylvania
  - Watson Investigational Site, Mountlake Terrace, Washington
  - Watson Investigational Site, Spokane, Washington

REFERENCES:
- [Derived] Nickel JC, O'Leary MP, Lepor H, Caramelli KE, Thomas H, Hill LA, Hoel GE. Silodosin for men with chronic prostatitis/chronic pelvic pain syndrome: results of a phase II multicenter, double-blind, placebo controlled study. J Urol. 2011 Jul;186(1):125-31. doi: 10.1016/j.juro.2011.03.028. Epub 2011 May 14. PMID 21571345

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Silodosin 4 mg | Silodosin 8 mg | Placebo
Started | 52 | 45 | 54
Completed | 43 | 31 | 41
Not Completed | 9 | 14 | 13
Not completed — Adverse Event | 4 | 6 | 3
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 4 | 2
Not completed — Lost to Follow-up | 2 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silodosin 4 mg | Silodosin 8 mg | Placebo | Total
Number analyzed (Participants) | 52 | 45 | 54 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 41 | 51 | 136
  >=65 years | 8 | 4 | 3 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 49.2 (13.34) | 46.7 (15.57) | 49.0 (11.62) | 48.4 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 52 | 45 | 54 | 151
Region of Enrollment [Number; unit: participants]
  United States | 52 | 45 | 54 | 151

OUTCOME MEASURES:

1. Primary Outcome: National Institutes of Health-Chronic Prostatitis Symptom Index (NIH-CPSI) Total Score.
Description: Change from baseline In NIH-CPSI at Week 12. Three separate domain scores are calculated as pain, urinary symptoms, and quality of life impact. NIH-CPSI total score uses a 0 to 43 scale; 0 best, 43 worse symptoms.
Time Frame: 12 weeks
Population: The number of participants for analysis is determined by Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Units on a 0 to 43 scale
Arm/Group | Silodosin 4 mg | Silodosin 8 mg | Placebo
Number analyzed (Participants) | 52 | 45 | 51
Units on a 0 to 43 scale
  Baseline NIH-CPSI Total Score | 26.0 (6.29) | 26.8 (5.94) | 27.9 (6.21)
  Chage from Baseline in NIH-CPSI at Week 12 | -12.1 (9.32) | -10.2 (8.84) | -8.5 (7.23)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Silodosin 4 mg | Silodosin 8 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/52 | 0/45 | 0/54
Other Adverse Events (participants affected / at risk) | 22/52 | 25/45 | 12/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silodosin 4 mg (N=52) | Silodosin 8 mg (N=45) | Placebo (N=54)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silodosin 4 mg (N=52) | Silodosin 8 mg (N=45) | Placebo (N=54)
Retrograde Ejaculation (Reproductive system and breast disorders) | 14 (15) | 18 (18) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5) | 4 (5)
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5) | 0 (0)
Sinusitis (Infections and infestations) | 3 (4) | 2 (2) | 0 (0)
Libido Decreased (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (3) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Neurogenic Bladder (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less